CLINICAL TRIAL: NCT05331053
Title: MicroRNA Activation of LOX-1 Mechanisms in Endometriosis
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID halting human subjects research and preliminary data from this proposal were used to submit an NIH grant. The NIH grant was funded and 3 other protocols were launched.
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, Lacy Alexander, Professor of Kinesiology, Physiology, Penn State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00009584
Record Dates: First submitted 2022-04-08; First posted 2022-04-15 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Endometriosis
Keywords: Skin blood flow; Cholesterol; Statin; Intradermal Microdialysis
MeSH Terms: conditions — Endometriosis | interventions — Atorvastatin

STUDY DESIGN:
Intervention Model Description: Only women with endometriosis will complete this study. Once consented and screened, each subject is asked to take Atorvastatin (Lipitor, 10mg/day) for seven days. Participants will undergo experimental testing before and after the seven day intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Atorvastatin (Experimental): Oral atorvastatin (Lipitor) therapy (10mg/day) for seven days.
  Atorvastatin acts as a systemic LOX inhibitor.
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — Simvastation acts as a systemic LOX inhibitor.

SUMMARY:
Endometriosis is a disorder that occurs in women. With endometriosis, tissue that should be found in the womb is found in sites outside of the womb. This disorder impairs the function of the cells that line the body's blood vessels (endothelium). The endothelium helps to control blood flow in healthy vessels. Women with this disorder have an increased risk for high blood pressure and high cholesterol. They have a higher risk for cardiovascular disease, too. With this study, we will learn how endometriosis impairs the lining of blood vessels and increases the risk for disease.

DETAILED DESCRIPTION:
Epidemiologic data demonstrate a clear association between endometriosis, reproductive risk factors, inflammation and cardiovascular (CV) risk. Circulating factors, Low-density lipoprotein (LDL) and oxidized LDL (oxLDL), are two of many biomarkers of cardiovascular and inflammatory disease of endometriosis. An important signaling mechanism through which circulating LDL and oxLDL act is the lectin-like oxidized LDL receptor (LOX-1). LOX-1 signal transduction functionally results in pronounced endothelial dysfunction, a hallmark of CV. We hypothesis that one factor mediating the elevated risk of cardiovascular disease in endometriosis is microRNA (miRNA) activation of LOX-1 receptor mechanisms.

Specific Aim 1. To test the hypothesis that LOX-1 receptor activation is increased leading to endothelial dysfunction in endometriosis.

Specific Aim 2. To test the hypothesis that decreased microRNAs (i.e. let7-a, let7-b, let7-g, MiR98, Mi590-p) are driving increased LOX-1 receptor expression and function in endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18 and 45 years with endometriosis (diagnosis by prior laparoscopy by subject's own physician <5 years prior, and reported by the subject to the researchers)

Exclusion Criteria:

* Use of nicotine-containing products (e.g. smoking, chewing tobacco, etc.)
* Diabetes (HbA1C .6.5%)
* BP>140/90
* Taking pharmacotherapy that could alter peripheral vascular control (e.g. insulin sensitizing, cardiovascular medications)
* Pregnancy
* Breastfeeding
* Taking illicit and/or recreational drugs
* Abnormal liver function
* Rash, skin disease, disorders of pigmentation, known skin allergies
* Diagnosed or suspected metabolic or cardiovascular disease
* Persistent unexplained elevations of serum transaminases
* Known allergy to latex or investigative substances

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All endometriosis patients had a confirmed diagnosis prior to enrollment via laparoscopy.
Pre-assignment Details: 6 enrolled
Groups:
- Atorvastatin: Oral atorvastatin (Lipitor) therapy (10mg/day) for seven days.
Period: Overall Study
Arm/Group | Atorvastatin
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin: Oral atorvastatin (Lipitor) therapy (10mg/day) for seven days.
  Atorvastatin acts as a systemic LOX inhibitor.
  Atorvastatin: Simvastation acts as a systemic LOX inhibitor.
Arm/Group | Atorvastatin
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Nitric Oxide Dependent Vasodilation in the Skin
Description: area under the curve of laser Doppler flux/mean arterial pressure * log acetylcholine (mol/L)
Time Frame: before and after intervention (7 days)
Population: A subset (n = 6) of endometriosis patients participated in a seven-day oral atorvastatin (Lipitor®) therapy (10 mg/day). These subjects returned to the laboratory on day 7, having taken the final dose that morning.
Measure: Mean (Standard Error); unit: flux/MAP*logAch(mol/L)
Arm/Group | Atorvastatin
Number analyzed (Participants) | 6
flux/MAP*logAch(mol/L) | 200 (80)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: other
Arm/Group | Atorvastatin
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/53/NCT05331053/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/53/NCT05331053/ICF_001.pdf